CLINICAL TRIAL: NCT00069108
Title: An Open-Label Randomized Phase III Study of Intermittent Oral Capecitabine in Combination With Intravenous Oxaliplatin (Q3W) ("XELOX") Versus Bolus and Continuous Infusion Fluorouracil/ Intravenous Leucovorin With Intravenous Oxaliplatin (Q2W) ("FOLFOX4") as Treatment for Patients With Metastatic Colorectal Cancer Who Have Received Prior Treatment With CPT-11 in Combination With 5-FU/LV as First Line Therapy
Brief Title: A Study of Xeloda (Capecitabine) in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO16967
Record Dates: First submitted 2003-09-15; First posted 2003-09-18 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Oxaliplatin; Capecitabine

ARMS (2):
- XELOX (Experimental): Participants received XELOX (oxaliplatin and capecitabine). Oxaliplatin was administered 130 mg/m^2 intravenous (IV) infusion over 2 hours (every 3 weeks [Day 1]) before the first dose of capecitabine. Capecitabine was administered orally within 30 minutes after the end of a meal (breakfast and dinner) at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2), with first dose the evening of Day 1 and last dose the morning of Day 15, given as intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) for up to 8 cycles (24-weeks).
  Interventions: Drug: Oxaliplatin; Drug: capecitabine [Xeloda]
- FOLFOX-4 (Active Comparator): Participants received FOLFOX-4 (combination of oxaliplatin, leucovorin [LV] and 5-fluorouracil [5-FU] combination). Oxaliplatin was administered as an 85 mg/m^2 IV infusion over 2 hours (on Day 1 only); with LV infusion as 200mg/m^2 over 2 hours followed by 5-FU, given as 400mg/m^2 bolus injection over 2-4 minutes, and then as a 600 mg/m^2 continuous infusion over 22 hours. On Day 2, Leucovorin 200 mg/m^2 (alone), followed by 5-FU 400 mg/m^2 bolus injection over 2-4 minutes, and 5-FU 600 mg/m^2 continuous infusion was repeated over 22 hours. It was (2-week cycles comprising 48 hours of infusion and 12 days of rest) for up to 12 cycles (24- weeks).
  Interventions: Drug: 5 FU; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5 FU — As prescribed, in 2 week cycles
  Arms: FOLFOX-4
Drug: Leucovorin — As prescribed, in 2 week cycles
  Arms: FOLFOX-4
Drug: Oxaliplatin — As prescribed, in 3 week cycles
  Arms: XELOX
Drug: Oxaliplatin — As prescribed, in 2 week cycles
  Arms: FOLFOX-4
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-15 of each 3 week cycle
  Arms: XELOX

SUMMARY:
This 2 arm study will assess the efficacy and safety of intermittent oral Xeloda, or iv fluorouracil/leucovorin, in combination with intravenous Eloxatin (oxaliplatin) in patients previously treated for metastatic colorectal cancer. Patients will be randomized to receive either 1)XELOX (Xeloda 1000mg/m2 po bid on days 1-15 + oxaliplatin) in 3 week cycles or 2) FOLFOX-4 (oxaliplatin + leucovorin + 5-FU in 2 week cycles. The anticipated time on study treatment is until disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* metastatic colorectal cancer;
* >=1 target lesion;
* failed first-line chemotherapy with 5-fluorouracil and irinotecan.

Exclusion Criteria:

* previous treatment with oxaliplatin;
* progressive or recurrent disease during or within 6 months of completion of first-line chemotherapy;
* >=1 previous chemotherapeutic agent or systemic anticancer regimen for metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2003-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- United States (8):
  - Bakersfield, California
  - Colorado Springs, Colorado
  - Washington D.C., District of Columbia
  - Terre Haute, Indiana
  - St Louis, Missouri
  - Billings, Montana
  - Nyack, New York
  - Dallas, Texas
- Belgium (4):
  - Brussels
  - Ghent
  - Kortrijk
  - Mont-godinne
- Canada (15):
  - Edmonton, Alberta
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Saint Catherines, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Weston, Ontario
  - Laval, Quebec
  - Lévis, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan
- Croatia (2):
  - Split
  - Zagreb
- Finland (2):
  - Tampere
  - Turku
- France (7):
  - Avignon
  - Bordeaux
  - Chambray-lès-Tours
  - Limoges
  - Nîmes
  - Pessac
  - Rouen
- Tübingen, Germany
- Greece (2):
  - Heraklion
  - Thessaloniki
- Israel (7):
  - Beersheba
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (4):
  - Bergamo
  - Cattolica
  - Rimini
  - Udine
- Poland (3):
  - Bialystok
  - Krakow
  - Warsaw
- San Juan, Puerto Rico
- Belgrade, Serbia
- Bratislava, Slovakia
- Ljubljana, Slovenia
- South Africa (5):
  - Cape Town
  - Durban
  - Pietermaritzburg
  - Port Elizabeth
  - Pretoria
- South Korea (2):
  - Buchun
  - Seoul
- Spain (4):
  - Barcelona
  - Leganés
  - Madrid
  - Palma de Mallorca
- Taiwan (3):
  - Kueishan
  - Tainan
  - Taipei
- United Kingdom (4):
  - Denbigh
  - Manchester
  - Merseyside
  - Preston

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 09 Jul 2003 to 31 Aug 2006 at 87 centers in 19 countries.
Groups:
- FOLFOX-4: Participants received FOLFOX-4 (combination of oxaliplatin, leucovorin [LV] and 5-fluorouracil [5-FU] combination). Oxaliplatin was administered as an 85 mg/m^2 IV infusion over 2 hours (on Day 1 only); with LV infusion as 200mg/m^2 over 2 hours followed by 5-FU, given as 400mg/m2 bolus injection over 2-4 minutes, and then as a 600 mg/m^2 continuous infusion over 22 hours. On Day 2, Leucovorin 200 mg/m^2 (alone), followed by 5-FU 400 mg/m^2 bolus injection over 2-4 minutes, and 5-FU 600 mg/m^2 continuous infusion was repeated over 22 hours. It was (2-week cycles comprising 48 hours of infusion and 12 days of rest) for up to 12 cycles (24- weeks).
Period: Overall Study
Arm/Group | XELOX | FOLFOX-4
Started | 313 | 314
Completed | 100 | 95
Not Completed | 213 | 219
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Adverse Event | 64 | 42
Not completed — Death | 6 | 6
Not completed — Administration | 15 | 4
Not completed — Insufficient therapy | 117 | 144
Not completed — Violation criteria | 1 | 4
Not completed — Refused treatment | 5 | 10

BASELINE CHARACTERISTICS:
Population: All participants with written informed consent who were randomized to one of the two study arms were included in the Intent-to-treat (ITT) population. Participants in this population were analyzed according to the arm to which they were randomized
Groups:
- XELOX: Participants received XELOX (oxaliplatin and capecitabine). Oxaliplatin was administered 130 mg/m^2 IV infusion over 2 hours (every 3 weeks [Day 1]) before the first dose of capecitabine. Capecitabine was administered orally within 30 minutes after the end of a meal (breakfast and dinner) at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2), with first dose the evening of Day 1 and last dose the morning of Day 15, given as intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) for up to 8 cycles (24-weeks).
- Total: Total of all reporting groups
Arm/Group | XELOX | FOLFOX-4 | Total
Number analyzed (Participants) | 313 | 314 | 627
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (9.91) | 59.7 (10.55) | 60.2 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 123 | 242
  Male | 194 | 191 | 385

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the day of documented disease progression or death from any cause. It was based on tumor assessments made according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0, wherein progressive disease (PD) was defined as at least a 20% increase in the sum of the longest diameter (LD) of the target lesions (TLs), taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more new lesions or unequivocal progression of existing non-target lesions. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment confirming that they had not progressed. Participants with no tumor assessments after baseline but who were still alive at the time of the clinical cut-off were censored at date of randomization
Time Frame: Up to 3 years
Population: The per protocol (PP) population included randomized participants who received at least one dose of capecitabine, 5-FU, or oxaliplatin, or who did not had a major violation of protocol inclusion or exclusion criteria assessments.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 251 | 252
days | 154 [140 to 175] | 168 [145 to 182]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin (1.30) was compared with the upper limit of the 95% confidence interval (CI) of the hazard ratio (HR, XELOX vs FOLFOX-4) in the population; p = 0.00584, Chi-squared; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.87 to 1.24] — The pre-specified non-inferiority margin (1.30) was compared with the upper limit of the 95% confidence interval (CI) of the hazard ratio (HR, XELOX vs FOLFOX-4) in the population

2. Secondary Outcome: Progression Free Survival Based on Independent Review Committee Assessment
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the day of documented disease progression or death from any cause. It was based on tumor assessments made according to the RECIST version 1.0, wherein PD was defined as at least a 20% increase in the sum of the LD of the TLs, taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more new lesions or unequivocal progression of existing non-TLs. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment confirming that they had not progressed. Participants with no tumor assessments after baseline but who were still alive at the time of the clinical cut-off were censored at date of randomization. This PFS evaluation was based on Independent Review Committee Assessment.
Time Frame: Up to 3 years
Population: PP population excluded randomized participants who did not receive at least one dose of Capecitabine, 5-FU, or Oxaliplatin, or who had a major violation of protocol inclusion or exclusion criteria.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 251 | 252
days | 168 [139 to 183] | 162 [141 to 179]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Non-Inferiority or Equivalence — While the study was not designed to demonstrate non-inferiority in PFS based on IRC assessments the pre-specified margin (1.30) was compared with the upper limit of the 95% confidence interval (CI) of the hazard ratio (HR, XELOX vs FOLFOX-4) in the population; p = 0.00223, Chi-squared; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.74 to 1.17] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression Free Survival Based on Treatment Analysis- Intent To Treat Population
Description: Progression free survival (PFS) is defined as the time from date of randomization to day of documented disease progression or death from any cause. It was based on tumor assessments made according to the RECIST version 1.0, wherein PD was defined as at least a 20% increase in the sum of LD of the TLs, taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more new lesions or unequivocal progression of existing non-TLs. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment confirming that they had not progressed. Participants with no tumor assessments after baseline but who were still alive at the time of the clinical cut-off were censored at date of randomization. PFS was analyzed using an on-treatment approach included only disease progression and death that occurred no later than 28 days after the last confirmed intake of study medication in the primary study treatment phase.
Time Frame: Up to 3 years
Population: All participants who were randomized to one of the two study arms were included in the Intent To Treat (ITT) population. Participants were analyzed according to the arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
days | 145 [137 to 169] | 152 [137 to 172]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.91 to 1.37]

4. Secondary Outcome: Progression Free Survival Based on Treatment Analysis- Per Population
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the day of documented disease progression or death from any cause. It was based on tumor assessments made according to the RECIST version 1.0, wherein PD was defined as at least a 20% increase in the sum of the LD of the TLs, taking as reference the smallest sum LD recorded since the treatment started or appearance of one or more new lesions or unequivocal progression of existing non-TLs. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment confirming that they had not progressed. Participants with no tumor assessments after baseline but who were still alive at the time of the clinical cut-off were censored at date of randomization
Time Frame: Up to 3 years
Population: The PP population included randomized participants who received at least one dose of Capecitabine, 5-FU, or Oxaliplatin, or who did not had a major violation of protocol inclusion or exclusion criteria assessments.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 251 | 252
days | 153 [139 to 172] | 164 [142 to 175]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.95 to 1.47]

5. Secondary Outcome: Best Overall Response, Investigators' Assessments
Description: Best overall response is best response recorded from start of treatment until disease progression/recurrence where responses include complete response (CR), partial response (PR), or stable disease (SD). CR was defined as disappearance of all TLs, non-TLs along with normalization of tumor marker level. PR is at least 30% decrease in sum of the LD of TLs, taking as reference baseline sum LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking reference of smallest sum LD since treatment started. It was dependent on achievement of measurement and confirmation criteria. BOR .i.e. CR or PR was confirmed by repeat assessments performed within 4 weeks. For SD, follow-up assessments had to meet the SD criteria at least once after study entry within 6 to 8 weeks.
Time Frame: Up to 3 years
Population: All participants who were randomized to one of the two study arms were included in the ITT population. Participants in this population were analyzed according to the arm to which they were randomized.
Measure: Number; unit: participants
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
participants
  Investigator Assessed, Responders | 63 | 55
  Investigator assessed-CR | 0 | 2
  Investigator assessed-PR | 63 | 53
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; p = 0.4028, Chi-squared — p-value is for difference between response rates; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.79 to 1.77]

6. Secondary Outcome: Best Overall Response, Independent Review Committee Assessment
Description: Best overall response is best response recorded from start of treatment until disease progression/recurrence where responses include CR, PR, or SD. CR was defined as disappearance of all TLs, non-TLs along with normalization of tumor marker level. PR is at least 30% decrease in sum of the LD of TLs, taking as reference baseline sum LD. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking reference of smallest sum LD since treatment started. It was dependent on achievement of measurement and confirmation criteria. BOR .i.e. CR or PR was confirmed by repeat assessments performed within 4 weeks, for SD, follow-up assessments had to meet the SD criteria at least once after study entry within 6 to 8 weeks. This PFS evaluation was based on Independent Review Committee Assessment.
Time Frame: Up to 3 years
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
participants
  IRC Assessed, Responders | 48 | 39
  IRC assessed-CR | 0 | 0
  IRC assessed-PR | 48 | 39
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; p = 0.2911, Chi-squared — p-value is for difference between response rates; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.81 to 2.01]

7. Secondary Outcome: Overall Survival
Description: Overall survival was measured as the time from the date of randomization to the date of death. Participant who were not reported to have died at the time of the analysis were censored using the date they were last known to be alive.
Time Frame: Up to 3 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
days | 363 [320 to 412] | 382 [323 to 418]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin (1.30) was compared with the upper limit of the 95% CI of the hazard ratio (HR, XELOX vs FOLFOX-4) in the population; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.87 to 1.23]

8. Secondary Outcome: Time To Response
Description: Time to response (TOR) (best response of CR or PR) was measured as the time from randomization to the first date on which the measurement criteria for CR or PR (whichever status was recorded first) were met. CR for TLs was defined as disappearance of all TLs and for non-TLs as disappearance of all non-TLs and normalization of tumor marker level. PR was defined as at least 30% decrease in the sum of the LD of TLs, taking as reference the baseline sum LD.
Time Frame: Up to 3 years
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
participants
  Week 1-6 | 13 | 11
  Week 7-12 | 26 | 23
  Week 13-18 | 22 | 18
  Week 19-24 | 2 | 3

9. Secondary Outcome: Duration Of Response
Description: Duration of response (DOR) is defined as the time when CR or PR was first met up to first date that PD or death is documented. CR is defined as disappearance of all TLs and non TLs, PR is defined as at least 30% decrease in the sum of the LD of TLs, taking as reference the baseline sum LD. PD was defined as at least a 20% increase in the sum of the LD of the TLs, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions for the TLs or the appearance of one or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Up to 3 years
Population: All participants who were randomized to one of the two study arms were included in the Intent-to-treat (ITT) population. Participants in this population were analyzed according to the arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 313 | 314
days | 169 [142 to 192] | 190 [161 to 206]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.79 to 1.68]

10. Secondary Outcome: Time To Treatment Failure
Description: Time to treatment failure was defined as the time from the date of randomization to the first occurrence of adverse event (AE), insufficient therapeutic response, death, failure to return, or refusing treatment/being uncooperative/withdrawing consent.
Time Frame: Up to 3 years
Population: All participants who were randomized and received at least one dose of capecitabine, 5-FU, or oxaliplatin were included in the safety population. The safety population was used for the analyses of all safety parameters.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 311 | 308
days | 125 [106 to 139] | 121.5 [101 to 137]
Statistical Analysis 1: Comparison: XELOX vs FOLFOX-4; Test type: Superiority or Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.81 to 1.12]

11. Secondary Outcome: Number of Participants With Marked Post-baseline Laboratory Abnormalities by Trial Treatment
Description: Laboratory abnormalities were defined as those values that were outside the Roche defined reference range and showed a clinically relevant change from baseline. All laboratory parameters were categorized according to the National Cancer Center Common Toxicity Criteria (NCI-CTCAE) grading system. Incidence of Grade 1 to 4 laboratory abnormalities are presented in the table below.
Time Frame: Up to 3 years
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | XELOX | FOLFOX-4
Number analyzed (Participants) | 311 | 308
participants
  Serum Glutamic-Pyruvic Transaminase (SGPT) | 90 | 110
  Serum Glutamic Oxaloacetic Transaminase (SGOT) | 193 | 174
  Alkaline Phosphatase | 184 | 201
  Calcium (hyper) | 7 | 9
  Calcium (hypo ) | 68 | 70
  Glucose (hyper) | 201 | 207
  Glucose (hypo) | 12 | 9
  Granulocytes | 1 | 6
  Haemoglobin | 216 | 240
  Neutrophils | 113 | 199
  Neutrophils/Granulocytes | 114 | 202
  Platelets | 168 | 212
  Potassium (hyper) | 17 | 26
  Potassium (hypo) | 68 | 92
  Serum Albumin | 116 | 138
  Serum Creatinine | 18 | 32
  Sodium (hyper) | 14 | 21
  Sodium (hypo) | 64 | 73
  Total Bilirubin | 107 | 95
  White blood cell (WBC) | 124 | 205

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who were randomized and received at least one dose of capecitabine, 5-FU, or oxaliplatin and had a safety assessment performed post baseline.
Arm/Group | XELOX | FOLFOX-4
Serious Adverse Events (participants affected / at risk) | 94/311 | 97/308
Other Adverse Events (participants affected / at risk) | 302/311 | 298/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX (N=311) | FOLFOX-4 (N=308)
Diarrhoea (Gastrointestinal disorders) | 18 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 8 | 4
Vomiting (Gastrointestinal disorders) | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Enteritis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
*Stomatitis all (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Infection (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 3
Abdominal abscess (Infections and infestations) | 0 | 2
Central line infection (Infections and infestations) | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 11
Neutropenia (Blood and lymphatic system disorders) | 0 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Warm type haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 9
Asthenia (General disorders) | 1 | 1
Catheter related complication (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Superior vena caval occlusionq (Vascular disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 5
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Analgesic therapy (Surgical and medical procedures) | 0 | 1
Urinary tract operation (Surgical and medical procedures) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX (N=311) | FOLFOX-4 (N=308)
Nausea (Gastrointestinal disorders) | 185 | 172
Diarrhoea (Gastrointestinal disorders) | 168 | 148
Vomiting (Gastrointestinal disorders) | 132 | 105
Abdominal pain (Gastrointestinal disorders) | 92 | 73
Stomatitis all (Gastrointestinal disorders) | 42 | 92
Constipation (Gastrointestinal disorders) | 50 | 79
Dyspepsia (Gastrointestinal disorders) | 34 | 23
Abdominal pain upper (Gastrointestinal disorders) | 20 | 18
Paraesthesia (Nervous system disorders) | 103 | 98
Peripheral sensory neuropathy (Nervous system disorders) | 40 | 50
Dysaesthesia (Nervous system disorders) | 32 | 34
Neuropathy peripheral (Nervous system disorders) | 40 | 30
Neuropathy (Nervous system disorders) | 36 | 29
Headache (Nervous system disorders) | 32 | 32
Hypoaesthesia (Nervous system disorders) | 23 | 20
Lethargy (Nervous system disorders) | 18 | 19
Dizziness (Nervous system disorders) | 32 | 29
Dysgeusia (Nervous system disorders) | 22 | 33
Fatigue (General disorders) | 127 | 129
Asthenia (General disorders) | 60 | 56
Pyrexia (General disorders) | 64 | 68
Temperature intolerance (General disorders) | 15 | 21
Oedema peripheral (General disorders) | 16 | 28
Chills (General disorders) | 9 | 18
Neutropenia (Blood and lymphatic system disorders) | 56 | 146
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 51
Anaemia (Blood and lymphatic system disorders) | 19 | 26
Anorexia (Metabolism and nutrition disorders) | 98 | 84
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 17
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 32 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 22
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 41
Pain in jaw (Musculoskeletal and connective tissue disorders) | 16 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 21
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 71 | 18
Rash (Skin and subcutaneous tissue disorders) | 30 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 19
Insomnia (Psychiatric disorders) | 21 | 37
Flushing (Vascular disorders) | 8 | 19
Weight decreased (Investigations) | 19 | 20
Nasopharyngitis (Infections and infestations) | 14 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.